CLINICAL TRIAL: NCT02484976
Title: Brain Systems and Behaviors Underlying Response to Obesity Treatment in Children
Brief Title: Brain Activation and Satiety in Children: Functional Magnetic Resonance Imaging
Acronym: BASIC-FMRI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Seattle Children's Hospital (Other)
Collaborators: University of Washington (Other)
Responsible Party: Principal Investigator, Christian Roth, Christian Roth, MD, Seattle Children's Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: R01DK098466 (NIH)
Record Dates: First submitted 2014-11-20; First posted 2015-06-30 (Estimated); Last update posted 2018-09-06 (Actual); Status verified 2018-09

CONDITIONS: Childhood Obesity
Keywords: Family Based Behavioral Treatment; functional magnetic resonance imaging (fMRI); Childhood Obesity; Satiety; BMI z-score; Impulsive; Non-obese controls; Visual food cues; Leptin; Hormones
MeSH Terms: conditions — Pediatric Obesity; Impulsive Behavior

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Family Based Behavioral Treatment (Experimental): Central satiety brain and hormonal responses will be compared pre-and post-Family Based Behavioral Treatment, as well, as to a non-obese sample.
  Interventions: Behavioral: Family Based Behavioral Treatment

INTERVENTIONS:
Behavioral: Family Based Behavioral Treatment — Obese children accompanied by at least one parent or caregiver will attend 24 weekly in-person sessions. Sessions will include 25-30 min. meetings between an interventionist and each child/parent pair to individualize treatment, followed by separate child and parent group meetings lasting 40 - 45 min. Parents will serve as primary agents of change for their child and for themselves. Training will focus on food and physical activity education, parenting around food and physical activity, and use of behavioral skills (e.g., self-monitoring, environmental control, contingency management). Intervention groups of 9-11 children/families will be initiated every 3-6 mos. in study yrs. 1-3.

SUMMARY:
BASIC fMRI is a prospective single center intervention trial using fMRI imaging in 9-11 year old obese male and females pre and post family-based behavioral treatment of 24 weeks duration to determine the relationship between impulsivity and central satiety responses.

DETAILED DESCRIPTION:
The high prevalence of childhood obesity in the U.S. demands a better understanding of factors that drive weight gain and influence the outcome of pediatric obesity interventions. This project investigates the hypothesis that, as in adults, a subset of obese children experience a diminished satiety response to food consumption, and that these children are more resistant to gold standard family-based behavioral treatment (FBT) for obesity. FBT is targeted almost exclusively toward parents; however, there is evidence that obesity development and response to intervention may depend on additional factors such as individual internal satiety perception and variability in the function of brain centers associated with impulsivity and reward. The proposed research uses functional magnetic resonance imaging (fMRI) to characterize brain function related to satiety and examines fMRI along with behavioral, cognitive, and hormonal testing to fully examine potential mediators of children's experience of satiety and response to FBT. The approach is based on evidence that failure to attenuate the reward value of palatable foods after eating can be a manifestation of a blunted central satiety response that is reliably detected using fMRI. Key objectives will be to determine if differences in the central satiety response exist between obese and non-obese children, and, among obese children, if the strength of the central satiety response is associated with impulsivity and/or the success of obesity treatment. The central hypothesis is that, in obese children, a blunted central nervous system satiety response impairs the success of obesity interventions. To achieve study objectives, brain activation by high-calorie visual food cues before and after food consumption will be measured by fMRI. Participants will be obese and non-obese children aged 9-11 years. The 49 obese children will be evaluated before and after they participate in a 6-month evidence-based FBT intervention. Their pre-intervention fMRI will be compared to those of 20 non-obese controls to test for a blunted central satiety response (Aim 1). The relationship of impulsivity to satiety responses and food intake will be determined in obese children (Aim 2). The longitudinal component tests whether central satiety responses prior to treatment predict treatment outcomes (Aim 3A) and whether changes in central satiety responses during treatment predict maintenance of reduced weight 6 and 12 months after treatment cessation (Aim 3B). Behavioral, cognitive, and hormonal measures will be examined as potential mediating or confounding factors contributing to fMRI responses. The proposed research is guided by an integrated, transdisciplinary team with expertise in pediatric and adult neuroimaging, appetite regulation, and family-based childhood obesity treatment. This research will provide new insights into the neurobiological basis of child obesity and the relevance of neurobiological factors to treatment success. The long-term objective is to translate these findings to improve obesity interventions cost-effectively and sustain better long-term results.

During years 1-3, obese children will be enrolled into intervention groups of 9-11 families with staggered start dates by 3-6 months. Years 1-4 includes enrollment, intervention, longitudinal follow-up, and data collection for obese children. Control children will primarily be recruited during years 2-3 to facilitate matching. FMRI scans are processed on a rolling basis as studies are completed. In years 3 and 4 hormonal assays will be performed. Final data analyses will be completed in year 4.

ELIGIBILITY:
Inclusion Criteria:

* 9-11 years of age
* Male or female
* Ability and willingness to participate in study visits including fMRI scans and blood draws;
* ability to provide informed written consent and assent;
* BMI z-score for lean control children 15th to 84.9th perc. for age and sex,
* BMI z-score for obese children BMI z-score >90th perc. for age and sex;
* Additional inclusion criteria for obese children: One overweight parent (BMI >25 kg/m2); willingness of 1 parent (does not have to be the obese parent) to engage in family-based weight control treatment.

Exclusion Criteria:

* History of acute or chronic serious medical conditions;
* known diabetes mellitus or recent (6 mo.) history of anemia;
* presence of any implanted metal or metal devices, including ferro-metallic surgical clips or braces;
* claustrophobia;
* documented cognitive disorder, disruptive behavior, inability to participate in group sessions;
* current use of medications known to alter appetite, body weight, or brain response (e.g. anti-seizure medications, glucocorticoids, medications for attention deficit disorder);
* food intolerance or vegetarianism.

Ages: 9 Years to 11 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 81 (Actual)
Dates: Start 2014-09; Primary Completion 2018-07 (Actual); Study Completion 2018-08 (Actual)

PRIMARY OUTCOMES:
Blunted central satiety response measured by functional magnetic resonance imaging | Baseline

SECONDARY OUTCOMES:
Change of brain response to visual food cues or eating behavior measured by functional magnetic resonance imaging | Change from pre- to post-treatment (end of 6 month intervention)
Relationship between impulsivity and satiety in obese children as measured by functional magnetic resonance imaging. | Change from pre- to post-treatment (end of 6 month intervention)
Relationship between impulsivity and satiety in obese children as measured by the Relative Reinforcing Value of Food (RRV). | Change from pre- to post-treatment (end of 6 month intervention)
Relationship between impulsivity and satiety in obese children as measured by the Developmental NEuroPSYchological Assessment (NEPSY). | Change from pre- to post-treatment (end of 6 month intervention)
Relationship between impulsivity and satiety in obese children as measured by the Delayed Choice Questionnaire (DCQ). | Change from pre- to post-treatment (end of 6 month intervention)

OTHER OUTCOMES:
Predictors of treatment outcomes measured by functional magnetic resonance imaging. | Change from pre- to post-treatment (end of 6 month intervention)
Predictors of treatment outcomes measured by behavioral skills use questionnaires. | Change from pre- to post-treatment (end of 6 month intervention)
Predictors of treatment outcomes measured by hormonal measures. | Change from pre- to post-treatment (end of 6 month intervention)

CONTACTS AND LOCATIONS:
Overall Officials: Christian Roth, MD, Principal Investigator — Seattle Children's Hospital
Locations (1):
- Seattle Childrens Hospital, Seattle, Washington, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Saelens BE, Melhorn SJ, Rowland MG, Scholz K, De Leon MRB, Elfers CT, Schur EA, Roth CL. General and Food-Specific Impulsivity and Inhibition Related to Weight Management. Child Obes. 2022 Mar;18(2):84-91. doi: 10.1089/chi.2021.0080. Epub 2021 Aug 5. PMID 34357785
- [Derived] Roth CL, Melhorn SJ, Elfers CT, Scholz K, De Leon MRB, Rowland M, Kearns S, Aylward E, Grabowski TJ, Saelens BE, Schur EA. Central Nervous System and Peripheral Hormone Responses to a Meal in Children. J Clin Endocrinol Metab. 2019 May 1;104(5):1471-1483. doi: 10.1210/jc.2018-01525. PMID 30418574